CLINICAL TRIAL: NCT03461549
Title: Open-label Preliminary Assessment of a Thin Flexible Pressure and Temperature Sensor for Therapeutic Compression Garments Using a Cohort of Healthy Adults Phase 2: Point-of-Care Wearable Pressure/Temp Sensor System for Therapeutic Compression Garments in Venous Leg Ulcers
Brief Title: Pressure and Temperature Sensor for Therapeutic Compression Garments
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Wearifi, Inc. (Unknown)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Instructor, Northwestern University
Other Study IDs: 090717SX
Record Dates: First submitted 2018-02-28; First posted 2018-03-12 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Healthy Adults; Venous Leg Ulcer
Keywords: pressure sensor; temperature sensor; wearables
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Healthy adults: Evaluate sensor performance on both lower limbs of healthy adult subjects for pressure sensing and skin temperature sensing.
  Interventions: Device: Pressure and Temperature Sensor
- Venous Leg Ulcer Adults: Evaluate sensor performance on both lower limbs of adult subjects with an active venous leg ulcer or history of a venous leg ulcer for pressure sensing and skin temperature sensing.
  Interventions: Device: Pressure and Temperature Sensor

INTERVENTIONS:
Device: Pressure and Temperature Sensor — This device includes pressure and temperature sensor embedded within silicone and applied to the skin with a medical grade adhesive.

SUMMARY:
Pilot study of a soft, flexible pressure and temperature sensor

DETAILED DESCRIPTION:
Assessment of safety, and preliminary accuracy of a pressure and temperature sensor adherent to the skin. The pressure sensor includes a piezoresistive fabric coupled to a near-field communication chip with a built-in temperature sensor.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults over the age of 18 years old

Exclusion Criteria:

* Subjects with history of medical or surgical problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults without a history of medical or surgical problem. There will be no subject compensation.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Pressure comparison with PicoPress | 72 hours
  Percent variation for each subject for pressure
Temperature with a comparator device (infrared camera) | 72 hours
  Percent variation for each subject for temperature

SECONDARY OUTCOMES:
Visual analogue scale of skin irritation | 72 hours
  A minimum score is 0 and a maximum score is 100 with a range of 0-100. A score of 0 is defined as no visible clinical appreciation. A score of 100 is defined as severe skin irritation. Higher values indicate worse outcome. There are no subscales.
Participant survey | 15 minutes
  Survey regarding the comfort of the sensor

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xu, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No